CLINICAL TRIAL: NCT06439186
Title: Infiltrative Anesthesia With Lidocaine Can Replace The Inferior Alveolar Nerve Block In Extraction of Devitalized Mandibular Molar Teeth
Brief Title: The Use of Infiltrative Anesthesia Instead of Inferior Alveolar Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Kubilay Isik, Professor, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KonyaNEU 2
Record Dates: First submitted 2024-05-02; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Local Infiltration
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthesia (Active Comparator): In the first group, inferior alveolar anesthesia is used. In the second group, infiltrative anesthesia is used.
  In both groups, one dose of lidocaine HCl contained in 2 mL ampule is used. It is a standard drug.
  Interventions: Drug: Lidocain
- tooth extraction pain (Active Comparator): In both groups, the patient is asked to evaluate the pain she/he experienced during the extraction. This evaluation is done immediately after the extraction, by using a "visual analogue scale" (detailed in other sections of this trial record).
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Lidocain — Local anesthesia
  Other Names: Lidocaine

SUMMARY:
Generally it is accepted that infiltrative anesthesia (IA) is not sufficient for extraction of lower molars and that an inferior alveolar nerve block (IANB) is needed. In this study, it was aimed to compare the effectiveness of IANB and IA in extraction of devitalized mandibular molars.

Sixty subjects are randomly divided into study (n=30) and control (n=30) groups. Lidocaine with epinephrine is used for all injections. In the study group only vestibular and lingual IA will be used. In the control group, IANB will be applied. Teeth were extracted as usual. The pain felt during extraction will be compared.

DETAILED DESCRIPTION:
It has been taught in dental curricula that using only infiltrative anesthesia (IA) is not sufficient for extraction of lower molars and that an inferior alveolar nerve block (IANB) is needed. However, it is also well-known that dental implants can be inserted into mandibular posterior region using only IA.

It can be claimed that there is no difference regarding the need for anesthesia between extracting a devitalized tooth and placing an implant in the same area. In this study, it was aimed to compare the effectiveness of IANB and IA in extraction of mandibular molars that had previously undergone root canal treatment.

The study is as a prospective, randomized, and non blinded clinical trial. All procedures are carried out at Necmettin Erbakan University, Faculty of Dentistry. The inclusion criteria are: age > 18 years, the tooth to be extracted is a mandibular first or second molar with a previously completed root canal treatment. The patients allergic to local anesthetics, those with severely mobile teeth, those had severe pain due to an acute infection, and the patients using psychotropic drugs are excluded.

Sixty subjects are randomly divided into study (n=30) and control (n=30) groups. An anesthetic solution containing 20 mg/mL of lidocaine and 0.0125 mg/mL of epinephrine was used in all subjects. In the study group only vestibular and lingual IA will be used. In the control group, IANB will be applied. The teeth will be extracted as usual. Using a visual analog scale (VAS), the pain felt during extraction will be separately recorded. Mann-Whitney U test will be used for statistical analysis. Statistical significance is defined as p<.05.

ELIGIBILITY:
Inclusion Criteria:

* the patient is older than 18 years
* the tooth to be extracted is a mandibular first or second molar with a previously completed root canal treatment

Exclusion Criteria:

* The patients allergic to local anesthetics
* Those with severely mobile teeth
* Those had severe pain due to an acute infection
* The patients using psychotropic drugs

Ages: 19 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Immediately after the tooth extraction.
  This is a 100 mm linear scale used to measure pain. On the left end is a description: "No pain at all. On the right end, there is the description "The worst pain imaginable." The patient will be asked to mark the pain on this line and then the distance from the left end to the mark will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Tunçdemir, PhD, Study Chair — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No